CLINICAL TRIAL: NCT02279199
Title: Assessment of Motor Proficiency in People With Bleeding Disorders Using the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2™)
Brief Title: Motor Proficiency of People With Bleeding Disorders Using the BOT-2 (TM)
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Oleson, Bethany Sloane DPT,PCS, Assistant Professor, Oregon Health and Science University
Other Study IDs: Motor Proficiency & Hemophilia
Record Dates: First submitted 2014-02-10; First posted 2014-10-31 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Hemophilia
Keywords: hemophilia; joint health; motor development; motor proficiency
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Normative data from standardized assessment
- Hemophilia: Persons aged 4-21 with any severity of hemophilia A or B

SUMMARY:
The purpose of this study is to find out if gross motor skills of children and young adults with bleeding disorders are different from those without bleeding disorders. The investigators will use the standardized motor test the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2 tm). The second purpose is to establish if history of joint disease secondary to bleeding affects gross motor skills.

1. Participants and setting: Subjects will include up to 100 male youth and young adults, ages 4 to 21, recruited from the patient population of the Hemophilia Treatment Center at OHSU. A mailing that describes the study may be sent to all potential subjects who receive care through the Hemophilia Treatment Center at OHSU. Data collection will occur at either clinic visits or in the home. Information, including history of change in joint structure and synovium, from existing bleeding disorder repositories at OHSU will also be used.
2. Design and Procedures: Research will be done using a prospective, cross-sectional study design to examine any relationship between a diagnosis of bleeding disorder and gross motor development. The gross motor ability of children and young adults with bleeding disorders who meet the inclusion criteria will be compared to sex-specific normative data from a standardized motor test. Information about age, type of hemophilia, presence of an inhibitor, type of management used, body composition, range of motion, and hand strength will also be collected through direct measurement and chart review. The information collected will be entered into a repository. A subject may choose to opt out of the repository while still participating in the research study. In addition, information from a current hemophilia repository will be compared to gross motor ability scores to determine if joint disease is related to skill level in this group of people.
3. Proposed analyses: Two-tailed t tests and logistic regression will be used to determine if there are any significant differences.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine whether gross motor proficiency of children and young adults with hemophilia falls below average, sex-specific normative data, using the standardized motor assessment the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2™). The primary hypothesis is that children and young adults with hemophilia perform at a lower level of gross motor proficiency compared to same-aged peers, despite advances in care.

The secondary purpose is to establish whether there is a relationship between joint health and level of gross motor proficiency. The secondary hypothesis is that history of hemophilia-caused ankle, knee, or elbow arthropathy will result in significant differences in gross motor proficiency within and between the populations of children and young adults with hemophilia.

Background/justification/rationale With the advent of widely-used prophylactic treatment for people with bleeding disorders, activity-limiting joint disease may be significantly reduced. Research investigating joint health and aerobic capacity of boys with hemophilia, an X-linked bleeding disorder, have shown no significantly different levels of functional ability when compared to peers, though other parameters may continue to be lower. However, a recent unpublished report of preliminary data using the Bruinicks-Oseretsky Test of Motor Proficiency (BOT-2 tm), a standardized gross motor assessment tool, suggests that male children and young adults with bleeding disorders function at a significantly lower level of gross motor skills compared to normative, sex-specific data, established when standardizing the BOT-2. This question is important in the determination of prognosis and intervention in this population.

Study Design Research will be conducted utilizing a prospective, cross-sectional study design to analyze the relationship between a diagnosis of bleeding disorder and gross motor development in male children and young adults as well as the association between joint health and gross motor development. As diagnosis of hemophilia is extremely rare in women and statistical analysis requires use of sex-specific normative data, this research study will focus strictly on the population of boys and young men with a diagnosis of hemophilia.

Once informed consent and assent (if applicable) is obtained, data will be collected by OHSU research personnel during a regular clinic visit at the Hemophilia Treatment Center (HTC). If a subject is unable to visit the clinic, informed consent/assent and study visit may be performed at the subject's home.

Recruitment Methods Potential subjects will be recruited during any clinic visit to the Hemophilia Treatment Center at OHSU. An IRB-approved recruitment letter may also be mailed to the Hemophilia Treatment Center's mailing list to recruit potential subjects.

Consent Process Informed, face-to-face consent will be sought prior to the collection of any data. Following a detailed explanation of the components of the study, the parent or legal guardian of the subject, if the subject is under 17, or the subject themselves may sign the informed consent. Assent will be obtained from patients aged 7-17. All children eligible for participation in the study and under the age of 17 will be assessed for their understanding prior to signing the assent form. Should the subject or their parents be non-English speaking, an in-person interpreter will be present for the entire consenting process to ensure understanding.

Study Procedures Data collection will take place in one clinic visit or one home visit by OHSU personnel. An interpreter will be scheduled should the family require an interpreter during a home visit or clinic visit. If data collection is not completed in one visit, a return visit, either to the clinic or to the home, will be conducted.

Clinical Data Current clinical data will be collected from the subject's medical record. Clinical data includes body composition recorded as Body Mass Index (BMI), type of bleeding disorder, severity, presence of inhibitor, method of management, and age. If a current height and weight is not available in the chart and the data collection occurs in the subject's home, appropriate devices for measurement of height and weight will be supplied to the investigators for this visit. This data will be transcribed onto the data collection sheet for each subject. Collected data will then be deposited into the data collection spreadsheet.

In addition, existing hemophilia repositories IRB # e5102 & IRB # e7074 will be accessed for each subject in the study to collect the following data: clinical joint health, as documented using the Hemophilia Joint Health Score (HJHS), and presence of chronic synovitis. Collected data will be deposited into the data collection spreadsheet.

Range of Motion During the subject's clinic or home visit, assessments of range of motion of hip flexion and extension, knee flexion and extension, ankle dorsiflexion and plantarflexion, elbow flexion and extension, forearm pronation and supination, and shoulder flexion will be taken using a goniometer and musculoskeletal landmarks according to standard clinical practice at the Hemophilia Treatment Center at OHSU.

Strength Subjects grip strength will be measured with hand held dynamometry. The Jamar Hydraulic Hand Dynamometer will be used to assess the bilateral grip strength in each subject, using the protocol set forth in the Jamar Owner's Manual.

Gross Motor Proficiency Gross motor proficiency will be assessed utilizing the following subtests of the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2™): Upper-Limb Coordination, Bilateral Coordination, Balance, Running Speed, and Agility and Strength. Prior to administration of the subtests, the researcher will determine the subject's hand and foot preferences for writing, throwing, and kicking, to be used within each subtest that requires use of a preferred extremity. Testing environment and test administration will conform to the protocol set out in the BOT-2™ Administration Manual.

ELIGIBILITY:
Inclusion Criteria:

* Patient of the Hemophilia Treatment Center at OHSU
* Male
* Aged 4 years, 0 months to 21 years, 11 months
* Diagnosis of bleeding disorder

Exclusion Criteria:

* Acute bleed or injury in the last two weeks that prevents activity
* Diagnosed developmental delay

Ages: 4 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and young adults with hemophilia A or hemophilia B, between the ages of 4 years, 0 months to 21 years, 11 months.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Motor Proficiency | At point of testing
  Motor proficiency of children and young adults with hemophilia compared to age-matched standardized norms

SECONDARY OUTCOMES:
Joint health using Hemophilia Joint Health Score (HJHS) | at point of testing
  Comparison of HJHS to standardized motor proficiency assessment to determine relationship between joint health and motor development

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Oregon Health and Science University, Portland, Oregon
  - Patient's home, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
There is a repository that is part of the consent process. Subjects can opt out if desired.
Supporting Information: Study Protocol, SAP
Time Frame: The manuscript is in progress. Once published, data will be available via the IRB approved repository if all conditions of the recipient IRB and the OHSU IRB are met.
Access Criteria: Approval of recipient and OHSU IRBs, respository guardian's approval.